CLINICAL TRIAL: NCT00902395
Title: Randomized Controlled Trial of Oral Sedatives for Moderate Sedation in Young Children
Brief Title: Efficacy of Moderate Sedation for Dental Treatment of Young Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Luciane Ribeiro de Rezende Sucasas da Costa, Associate Professor, Faculty of Dentistry, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFG SAP 18189
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Dental Caries; Child Behavior; Conscious Sedation Failure During Procedure
Keywords: Preschool children
MeSH Terms: conditions — Dental Caries; Child Behavior | interventions — Midazolam; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midazolam (Active Comparator): Oral midazolam
  Interventions: Drug: Midazolam
- Midazolam/ketamine (Experimental): Combined midazolam and ketamine
  Interventions: Drug: Midazolam, ketamine
- Protective stabilization (Other): No drug or placebo administered
  Interventions: Behavioral: Protective stabilization

INTERVENTIONS:
Drug: Midazolam — Oral midazolam 1.0 mg/kg (maximum 20 mg)
  Other Names: Dormire, Cristalia, Sao Paulo, Brazil
  Arms: Midazolam
Behavioral: Protective stabilization — Children will receive a protective stabilization (physical restrain) with sheet fixed with tapes.
  Other Names: No drug administered
  Arms: Protective stabilization
Drug: Midazolam, ketamine — Combined oral midazolam (0.5 mg/kg) and ketamine (3 mg/kg) (MK)
  Other Names: Dormire, Cristalia, Sao Paulo, Brazil; Ketamin S+, Cristalia, Sao Paulo, Brazil
  Arms: Midazolam/ketamine

SUMMARY:
There is lack of clinical trials on pediatric dental sedation. The purpose of this study is to test (using a randomized controlled trial design) the hypothesis that young children behavior during dental treatment improves with oral midazolam sedation. A further aim of this study was is explore whether behavior also changes over sessions needed to dental treatment completion.

DETAILED DESCRIPTION:
There is a lack of clinical trials on pediatric dental sedation in children 3 years old and under. We investigated whether young children's behavior improves during dental treatment with combined oral ketamine and midazolam compared to midazolam alone or no sedation. Healthy children under 36 months of age, presenting early childhood caries and referred to a pediatric dental sedation clinic were randomly assigned to receive combined midazolam (0.5 mg/kg) and ketamine (3 mg/kg) (MK), oral midazolam (1.0 mg/kg) (MS), or protective stabilization without sedative (PS). One observer scored children's behavior using the Ohio State University Behavior Rating Scale (OSUBRS) at determined points in a dental exam (no sedative) and treatment session. Data were analyzed using non-parametric bivariate tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA PS 1)
* Children under 36 months old
* Children presenting early childhood caries
* Children with no history of dental treatment

Exclusion criteria:

* Lost to follow-up

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Children's behavior at the dental office after they had dental rehabilitation of early childhood caries when they were under 3 years old | 2 years

SECONDARY OUTCOMES:
Efficacy of oral sedation with midazolam during children's dental treatment comparing to protective stabilization | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Luciane R Costa, DDS, MS, PhD, Principal Investigator — Faculty of Dentistry, Federal University of Goias; Paulo S Sucasas, MD, MS, PhD, Principal Investigator — Medical School, Federal University of Goias; Thiago A C Moreira, MD, Study Chair — Health Sciences Graduate Program, UFG; Denise E Antunes, DDS, PhD, Study Chair — Health Sciences Graduate Program, UFG; Cristiana M Jesus-Franca, DDS, PhD, Study Chair — Health Sciences Graduate Program, UFG; Hugo S G Oliveira, MD, Study Chair — Health Sciences Graduate Program, UFG; Onofre A Neto, MD, PhD, Study Chair — Faculty of Medicine, UFG
Locations (1):
- Dental School, Goiânia, Goiás, Brazil

REFERENCES:
- [Result] Moreira TA, Costa PS, Costa LR, Jesus-Franca CM, Antunes DE, Gomes HS, Neto OA. Combined oral midazolam-ketamine better than midazolam alone for sedation of young children: a randomized controlled trial. Int J Paediatr Dent. 2013 May;23(3):207-15. doi: 10.1111/j.1365-263X.2012.01246.x. Epub 2012 May 28. PMID 22631626